CLINICAL TRIAL: NCT04088201
Title: Epidermal Adhesive Sensors to Enhance Continuous Glucose Measurement in Patients With Diabetes: The EASE Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Edward Chao, Clinical Professor of Medicine, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 190708
Record Dates: First submitted 2019-09-09; First posted 2019-09-12 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Measuring glucose (Experimental): Measuring glucose from interstitial fluid
  Interventions: Device: Glucose measurements

INTERVENTIONS:
Device: Glucose measurements — We will not conduct an intervention, but will obtain measurements from a continuous, non-invasive glucose sensor, and compare with those from a glucometer.

SUMMARY:
Self-testing of glucose by patients living with diabetes mellitus (DM) involves needles, which can cause discomfort or inconvenience; these and other factors can lead to decreased willingness to perform these checks that are vital to DM management. While technology has evolved, a needle-free glucose monitoring device is currently not available. The investigators are studying a glucose sensor that adheres to the skin, similarly to a temporary tattoo. This sensor can now obtain continuous readings. As it has not yet been tested in individuals with DM, this study will examine its accuracy and acceptability in these patients. Results from this clinical trial could serve as the basis for further development of a non-invasive, wearable glucose sensor that can provide measurements of glucose levels continuously.

ELIGIBILITY:
Inclusion Criteria:

* An existing diagnosis of diabetes mellitus, either T1DM or T2DM, or any other type or etiology of diabetes
* Ability to provide informed consent for participation.

Exclusion Criteria:

* Individuals without diabetes
* Those who cannot speak or read English. We are limiting participation to those who read and speak English, as this is a pilot study of a small number of participants, that will very unlikely offer the prospect of direct benefit from participating.
* Individuals who have frequent hypoglycemia, hypoglycemia unawareness, or who are at high risk for hypoglycemia.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-09-26 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Interstitial fluid glucose readings | Hourly, up to 8 hours
  Needle-less measurements with an epidermal sensor - pls note, study is to assess how sensor readings compare with those from a glucometer

SECONDARY OUTCOMES:
Acceptablility of sensor | At end of study testing sessions, at 8 hours
  Will survey pts

CONTACTS AND LOCATIONS:
Overall Officials: Edward C Chao, DO, Principal Investigator — UCSD
Locations (1):
- University of California, San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://cws.ucsd.edu/research